CLINICAL TRIAL: NCT05917210
Title: Peer-led Implementation of TB-HIV Education and Adherence Counseling in Uganda
Acronym: TEACH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2000035416; 1R01HL170926-01A1 (Other Grant/Funding Number: NIH)
Record Dates: First submitted 2023-06-14; First posted 2023-06-23 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Tuberculosis; HIV
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peer navigation strategy for TB Education and Counseling (TB-EC) (Experimental): peer-navigation strategy for TB-EC in adults and adolescents with and without HIV starting TB treatment at clinics in Uganda
  Interventions: Behavioral: Peer navigation strategy for TB-EC
- Standard TB-EC (Active Comparator): standard TB-EC in adults and adolescents with and without HIV starting TB treatment at clinics in Uganda
  Interventions: Behavioral: Standard TB-EC

INTERVENTIONS:
Behavioral: Standard TB-EC — Standard TB-EC by healthcare workers
  Arms: Standard TB-EC
Behavioral: Peer navigation strategy for TB-EC — multi-component, peer-navigation strategy for TB-EC
  Arms: Peer navigation strategy for TB Education and Counseling (TB-EC)

SUMMARY:
This cluster-randomized trial in Uganda will evaluate the effectiveness and implementation of a novel, peer-led TB education and counseling strategy to improve outcomes among persons with tuberculosis (TB) with and without HIV/AIDS and assess the social-behavioral mechanisms underlying the observed treatment effects.

DETAILED DESCRIPTION:
Study Design Aim 1. The investigators will conduct a parallel cluster-randomized hybrid Type 2 effectiveness-implementation trial at 16 sites.

Aim 2. Within the Aim 1 study, the investigators will nest a longitudinal observational study in both arms of the cluster-randomized trial to determine the feasibility, acceptability, and appropriateness of a peer-navigation strategy for TB-EC. The investigators will concurrently assess biological adherence using urine biomarkers) and will also perform a mediation analysis of social and behavioral factors (i.e., TB knowledge, perceived social support, general self-efficacy, HIV/TB stigma) to identify causal mechanisms of impact. Finally, the investigators will pilot and culturally adapt study instruments in a pilot study prior to the trial.

Aim 3. The investigators will also conduct a qualitative and mixed methods studies to assess the implementation fidelity and context of the peer-navigation strategy for TB-EC:

1. Process evaluation of intervention fidelity to quantify the adoption, reach, implementation, and maintenance of the peer navigation strategy,
2. In-depth interviews with people with Tuberculosis (PWTB) with and without HIV,
3. In-depth interviews with and direct observation of peer navigators, and
4. Focus-group discussions (FGDs) with healthcare workers.

The focus of this registration is Aim 1 and 2.

ELIGIBILITY:
Inclusion Criteria:

TB outcomes:

* Sites will enroll consecutive adults and older adolescents (age ≥18) recorded as new TB cases in the on-site National TB Program TB treatment register.

ART outcomes:

* Participants must be documented as a People Living with HIV (PLH) in the TB register.

Exclusion Criteria:

TB outcomes: Individuals who are

* transferring in from off-site
* diagnosed with possible or confirmed drug-resistant TB
* residing >40 km from the clinic
* lacking mental capacity to participate in peer counseling

will be excluded from this study.

ART outcomes:

* The investigators will exclude those with TB meningitis or TB pericarditis for which immediate ART is contraindicated; and those with central nervous system TB or TB osteomyelitis because these forms of TB have a different treatment duration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1920 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2027-11-30 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Effectiveness assessed by TB treatment completion | up to 8 months post TB treatment initiation
  The number of participants with TB treatment completion, defined by WHO as attending all refill visits and completing 180 daily doses of standard TB treatment within 8 months of TB treatment initiation, as documented in the on-site TB treatment register.
Effectiveness assessed by Antiretroviral Therapy (ART) retention | month 12 post ART initiation
  The number of participants with ART retention, defined as completing all ART refill visits (or refill pickups if enrolled in differentiated models of ART care) and continuing on daily ART 12 months after starting ART, as documented in the on-site ART register.

SECONDARY OUTCOMES:
Clinical Effectiveness assessed by TB recurrence-free survival | month 6 post TB-treatment
  Clinical Effectiveness assessed by the number of participants with 6-month post-treatment TB recurrence-free survival. Data collectors at all sites will telephone participants and/or treatment supporters to document TB recurrence-free survival.
Clinical Effectiveness assessed by HIV RNA copy number | month 12 post ART initiation
  Clinical Effectiveness assessed by the number of participants with 12-month HIV RNA ≤50 copies/mL.

CONTACTS AND LOCATIONS:
Overall Officials: J. Lucian Davis, MD, Principal Investigator — Yale University
Locations (1):
- Primary Care Clinics, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual data will be available on a public registry.